CLINICAL TRIAL: NCT03044184
Title: Randomized, Double-blind, Placebo-controlled Trial to Investigate the Effectiveness of Early Intravenous Tranexamic Acid in Limiting Hematoma Expansion in Patients With Spontaneous Intracerebral Hemorrhage
Brief Title: Tranexamic Acid for Spontaneous Acute Cerebral Hemorrhage Trial
Acronym: TRANSACT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Peter Woo Yat Ming, Doctor, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KwongWH
Record Dates: First submitted 2017-01-26; First posted 2017-02-06 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Stroke Hemorrhagic; Intracerebral Haemorrhage
Keywords: Tranexamic Acid; Antifibrinolytic
MeSH Terms: conditions — Hemorrhagic Stroke; Cerebral Hemorrhage | interventions — Tranexamic Acid; Tranylcypromine

STUDY DESIGN:
Intervention Model Description: Randomised placebo-controlled parallel group clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Intravenous normal saline or transamine will be administered to subjects. Both will be of equal volume, colour and in similar intravenous fluid packaging.
  The outcomes assessor will be unaware of the subject group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Standard management for patients with spontaneous intracerebral hemorrhage according to 2015 AHA/ASA Guidelines for the Management of Intracerebral Hemorrhage
  AND
  Patients will have 1gram of tranexamic acid (diluted in 100ml of normal saline 0.9%) intravenously infused over 10 minutes within 3 hours of symptom presentation and another 1 gram of tranexamic acid (diluted in 100ml of normal saline 0.9%) infused over 8 hours.
  Interventions: Drug: Tranexamic Acid
- Control (No Intervention): Standard management for patients with spontaneous intracerebral hemorrhage according to 2015 AHA/ASA Guidelines for the Management of Intracerebral Hemorrhage
  AND
  Patients will 100ml of normal saline 0.9% intravenously infused over 10 minutes within 3 hours of symptom presentation and another 100ml of normal saline 0.9% infused over 8 hours.

INTERVENTIONS:
Drug: Tranexamic Acid — Transamine is an antifibrinolytic medication given systemically via the intravenous route
  Other Names: Transamine
  Arms: Intervention

SUMMARY:
This study aims to explore the effectiveness of tranexamic acid (also known as trans amine or TXA) in reducing hematoma expansion in patients with hemorrhagic stroke when given in the acute phase.

METHODOLOGY

This will be a Phase III, parallel-group double-blind randomised placebo control trial. Patients allocated to the control group will receive standard care for hemorrhagic stroke according to the 2015 American Heart Association guidelines. Patients allocated to the intervention group will receive, in addition to standard care, a loading dose of intravenous TXA 1gm within 3 hours of symptom onset followed by a 1gm maintenance dose over 8 hours. Timing and dosing are in accordance to previous established study protocols. Patients in the intervention group will only receive a single treatment course of TXA.

Study subjects will be identified by either the on-duty clinicians from the Department of Neurosurgery of this institution or by the study investigators. Should the patient meet study eligibility criteria consent will be obtained either from the patient or from his/her next of kin. 1:1 block randomization will be performed by a remote internet randomization service by accessing a website. Patients allocated to the intervention arm will have 1gm of TXA added to 100ml of normal saline (0.9%) infused over 10 minutes as a loading dose. This is then followed by a maintenance dose of 1gm of TXA in 500ml of intravenous isotonic solution infused at 120mg/hour (60ml/hour) for 8 hours. Patient's allocated to the control arm will have an equal volume of normal saline (0.9%) infused as a placebo. The patient and the outcome assessor will be blinded to study group allocation.

The primary endpoint of this study will be to assess the percentage change in brain blood clot volume by computed tomography brain scans on admission, 6 hours later, at 24 hours and at 1 week.

DETAILED DESCRIPTION:
INTRODUCTION

There are very few treatment options for patients with spontaneous intracerebral hemorrhage, a type of hemorrhagic stroke especially prevalent among Chinese, during the acute phase. Blood clot expansion in the brain (hematoma expansion; HE) is one of the most significant predictors for poor outcome in such patients.

Tranexamic acid (TXA) is a commonly used medication available in all acute Hospital Authority hospitals prescribed for a variety of conditions when bleeding occurs, for example epistaxis and menorrhagia. Intravenous administration of TXA has been proven to benefit severe trauma patients by reducing mortality and also preventing the recurrent rupture of brain aneurysms in another type of hemorrhagic stroke. The medication is safe and has been proven to improve outcomes in these patients.

A previously performed pilot study exploring the safety and feasibility of administrating intravenous TXA to patients with hemorrhagic stroke was recently performed and concluded the medication's safety. There was also a trend to significance for reducing the percentage change of hematoma volume in patients who received TXA.

This study aims to explore the effectiveness of TXA in reducing hematoma expansion in patients with hemorrhagic stroke when given in the acute phase.

METHODOLOGY

This will be a Phase III, parallel-group double-blind randomised placebo control trial. Patients allocated to the control group will receive standard care for hemorrhagic stroke according to the 2015 American Heart Association guidelines. Patients allocated to the intervention group will receive, in addition to standard care, a loading dose of intravenous TXA 1gm within 3 hours of symptom onset followed by a 1gm maintenance dose over 8 hours. Timing and dosing are in accordance to previous established study protocols. Patients in the intervention group will only receive a single treatment course of TXA.

Study subjects will be identified by either the on-duty clinicians from the Department of Neurosurgery of this institution or by the study investigators. Should the patient meet study eligibility criteria consent will be obtained either from the patient or from his/her next of kin. 1:1 block randomization will be performed by a remote internet randomization service by accessing a website. Patients allocated to the intervention arm will have 1gm of TXA added to 100ml of normal saline (0.9%) infused over 10 minutes as a loading dose. This is then followed by a maintenance dose of 1gm of TXA in 500ml of intravenous isotonic solution infused at 120mh/hour (60ml/hour) for 8 hours. Patient's allocated to the control arm will have an equal volume of isotonic solution infused as a placebo. The patient and the outcome assessor will be blinded to study group allocation.

The primary endpoint of this study will be to assess the percentage change in brain blood clot volume by computed tomography brain scans on admission, 6 hours later, at 24 hours and at 1 week. Volumetric analysis of the brain scans will be performed by two radiologists blinded to the patient's study group allocation..

Secondary endpoints will be assessed by a research assistant blinded to the patient's study group allocation. One such endpoint is functional outcome in terms of the Glasgow Outcome Scale and modified Rankin scale at 3 months and 6 months after stroke. Another secondary endpoint is quality of life at 3 months and 6 months by adopting the Stroke-specific Quality of Life Scale. Other secondary endpoints include death within 30 days of admission, vascular occlusive events (myocardial infarction, pulmonary embolism, deep vein thrombosis), ischemic stroke, seizures and other TXA-associated adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CT evidence of supratentorial intracerebral hemorrhage
2. Initiation of trial medication within 3 hours from the time of symptoms onset.
3. Ethnic Chinese
4. Reasonable expectation of completion of outcome measures at follow-up
5. Written informed consent from either the patient or next-of-kin or legal guardian.

Exclusion Criteria:

1. Patients not expected to survive 24 hours after admission.
2. Patients with brainstem herniation syndrome on admission.
3. Patients who need immediate neurosurgical intervention.
4. GCS of of 5 or less on admission i.e. a GCS score of 2 according to the Hemphil ICH score1.
5. Previous antiplatelet and anticoagulant medication use.
6. Known thrombocytopenia or coagulopathy.
7. Disseminated intravascular coagulation on admission.
8. Acute sepsis on admission.
9. Intracerebral hemorrhage (ICH) secondary to intracranial vascular lesion: aneurysm, arteriovenous malformation, neoplasm or dural venous sinus thrombosis.
10. Previous venous thromboembolic disease : deep venous thrombosis.
11. History of ischemic stroke or transient ischemic attack within 12 months.
12. History of ischemic heart disease or myocardial infarction.
13. History of peripheral vascular disease.
14. Patients with previous disability (prestroke modified Rankin scale score >2)
15. Pregnancy or breast feeding.
16. History of allergy to tranexamic acid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracerebral hematoma volume (by computed tomography brain scan) at 6 hours | At 6 hours
  Intracerebral hematoma volume (ml) as assessed by CT brain scan.
Intracerebral hematoma volume (by computed tomography brain scan) at 24 hours | At 24 hours
  Intracerebral hematoma volume (ml) as assessed by CT brain scan.
Intracerebral hematoma volume (by computed tomography brain scan) at 1 week | At 1 week
  Intracerebral hematoma volume (ml) as assessed by CT brain scan.

SECONDARY OUTCOMES:
Glasgow outcome score | At 3-months and 6 months after stroke
Modified Rankin score | At 3-months and 6 months after stroke
Stroke-specific quality of life scale | At 3-months and 6 months after stroke
30-day mortality | At 30 days after admission or until time of death within 30 days
  All-cause mortality within 30 days of admission
Vascular occlusive events | At 30 days after admission
  Ischemic stroke, myocardial infarction, pulmonary embolism, deep vein thrombosis
Rate of seizures | At 30 days after stroke
  Rate of seizures within 30 days of stroke
Tranexamic acid-associated adverse effects | At 30 days after admission
  1. Intolerable gastrointestinal symptoms such as dyspepsia, diarrhea, vomiting.
  2. Allergic reaction to TXA.
Need for neurosurgical intervention | At 30 days after admission
  Need for operative management of the hemorrhagic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Peter YM Woo, FRCS, Principal Investigator — Neurosurgery, Kwong Wah Hospital
Locations (1):
- Kwong Wah Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112